CLINICAL TRIAL: NCT01627184
Title: Long-term Use: CGM System Assessment in Adult Athletes With Diabetes Mellitus
Acronym: LUCID
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-900905
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Athletes with diabetes mellitus: Athletes who are insulin-requiring and insulin-dependent diabetics undergoing high levels of activity over extended period of time
  Interventions: Device: Dexcom G4 CGM System

INTERVENTIONS:
Device: Dexcom G4 CGM System

SUMMARY:
The purpose of this study is to evaluate CGM glycemic control using the Dexcom G4 system as well as system performance during high levels of activity and home use by adult athletes with insulin-requiring diabetes mellitus, over an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of diabetes mellitus

Exclusion Criteria:

1. Extensive skin changes/diseases
2. Known allergy to medical adhesives
3. Pregnancy
4. Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult athletes with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Glycemic Control during Exercise | multiple months, up to 6
  The proportion of time spent in euglycemia zone as well as hypoglycemia zone will be determined from the system glucose readings, particularly during subject's high levels of activity. Longitudinal data analysis methods will be used to assess the within-subject and between-subject effects of the glycemic control for the study population.

SECONDARY OUTCOMES:
System Utility and Usability | multiple months, up to 6
  The objectives of the study are to evaluate the Dexcom G4 system utility and usability during high levels of activity and home use. The assessments may be evaluated by, but are not limited to, the following:
  * Number and duration of sensors used by subject
  * Percentage of CGM system communication during wear
  * Percentage of CGM system glucose reading during wear
  * Incidence of System prompts and error messages recorded in the receiver

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta Diabetes Association, Atlanta, Georgia, United States